CLINICAL TRIAL: NCT01251627
Title: A Phase II Multicenter Open-label Study to Assess the Efficacy of Decitabine in the Treatment of Chronic Myelomonocytic Leukemia
Brief Title: Multicenter Study to Assess the Efficacy of Decitabine in the Treatment of Chronic Myelomonocytic Leukemia
Acronym: DECI2009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DECI2009-AISSM06
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, Decitabine
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine (Experimental): Eligible patients will recieve Dacogen 20mg/m2 in 1 hour iv infusion for 5 days every 28 days (1 cycle)plus Best Supportive Care.A total of 6 courses is planned.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Decitabine will be administered at a dose of 20 mg/m2 infused over a 1 hour period once daily for 5 consecutive days. The totale amount per course is 100 mg/m2. Cycles will be administered every 4 weeks (1 cycle of 28 days).It is recommented that patients be treated for a minimum of 4 cycles.

SUMMARY:
The study aims to assess the activity of decitabine in the treatment of CMML.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and older
2. CMML diagnosis according to WHO criteria
3. If WBC<=12000/mm3:IPSS High or INT-2

   If WBC>12000/mm3: at least two of the following criteria:
   * Blast cells>5% in the bone marrow
   * Citogenetic abnormality other then t(5;12) (q33;p13)
   * Anemia (Hb<10g/dl)
   * Thrombocytopenia (Plt<100000/mm3)
   * Splenomegaly(>5cm below costal margin)
   * Extramedullary localization
4. Patients untretaed or previously treated with Hydroxyurea or Imatinib or Etoposide given orally or non intensive chemotherapy or intensive chemotherapy given more thann 3 months befor inclusion
5. Performance Status ECOG 0,1 or 2
6. Estimated life expectancy>=6 months
7. Adequate hepatic function:

   * Total bilirubin < 1.5 times upper limit of normal (except moderate unconjugate hyperbilirubinemia due to intra medullary hemolysis)
   * AST and ALT < 3 times limit of normal
8. Adequate renal function:

   * Serum creatinine < 1.5 times limit of normal
   * Creatinine clearance > 30ml/min
9. Informed consent
10. Negative pregnancy test or adequate contraception methods

Exclusion Criteria:

1. Myeloproliferative/myelodisplastic syndome othe than CMML
2. Acute blastic transformation of CMML with bone marrow blast cells>20%
3. Patients eligible for allogenic bone marrow transplantation with identified donor
4. CMML with t(5;12) o PDGFBR rearrangement
5. Intensive chemotherapy given less than 3 months before
6. Previous treatment with hypomethylating agent
7. Age< 18 years old
8. Pregnancy or breastfeeding
9. Performance Status ECOG>2
10. Estimate life expectancy<6 months
11. HIV infection
12. Chronic active hepatitis secondary to HCV or HBV (HBSAq positive)
13. Serious concomitantsystemic disorders, including active bacterial fungal or viral infection, that in the opinion of the investigator, would compromise the safety of the patient and/or his/her ability to complete the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
To assess the activity of decitabine in the treatment of CMML | 24 months
  Activity will be evaluated as percentage of patients achieving complete or partial remission according to the International Working Group response criteria in myelodysplasia

SECONDARY OUTCOMES:
to assess the activity of decitabine in the treatment of CMML in terms of overall survival, time to leukemic transormation, response duration in terms of time to relapse after CR, PR, time to disease progression, ecc | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Santini Valeria, Professor, Principal Investigator — U.O di Ematologia, AO of Careggi, viale Morgagni n.85-50134-Firenze
Locations (21):
- Italy (21):
  - Ematologia, Ospedale SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - AOU Ospedali Riuniti di Ancona, Ancona
  - Ematologia AOU Policlinico di Bari, Bari
  - Istituto di Ematologia e Oncologia Medica, Policlinico S.Orsola, Bologna
  - Ematologia - Spedali Civili, Brescia
  - Ematologia- Ospedale Businco, Cagliari
  - Centro di ricerca e formazione ad alta tecnologia nelle Scienze, Università Cattolica, Campobasso
  - Cattedra di Ematologia Policlino Careggi, Florence
  - Dipartimento Emato-Oncologia AOU San Martino Genova, Genova
  - Fondazione IRCCS Caà Granda-Ospedale Maggiore policlinico, Milan
  - Divisione di Ematologia, Ospedale S.Gerardo di Monza, Monza
  - Divisione di Ematologia, Università Avogadro, Novara
  - Medicina interna II Divisione di Ematologia Ospedale S.Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale S.Maria della Misericordia, Perugia
  - AOU San Salvatore, Pesaro
  - AO Bianchi Melacrino Morelli, Reggio Calabria
  - IRCCS Centri di riferimento oncologico, Rionero in Vulture
  - SC Ematologia AOU S.Andrea, Roma
  - Ematologia 2-Ospedale S.Giovanni Battista, Torino
  - U.O.Ematologia 2, Torino